CLINICAL TRIAL: NCT00270257
Title: A Phase III Randomized Controlled Trial to Evaluate the Efficacy of Drug Treatment in Prevention of HIV Infection and Death Among Opiate Dependent Injectors
Brief Title: Drug Treatment Combined With Drug and Risk Reduction Counseling to Prevent of HIV Infection and Death Among Injection Drug Users
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB halted the study due to futility as a result of lower than anticipated HIV incidence rates
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 058; 10144 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2016-12

CONDITIONS: HIV Infections; Opioid-Related Disorders
Keywords: HIV Seronegativity; Opiate Addiction; Opiate Dependence
MeSH Terms: conditions — HIV Infections; Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long term medication assisted treatment (LT-MAT) (Experimental): Participants will receive BUP/NX under the tongue daily for a maximum of three weeks(until dose stabilization) and then three times a week for 52 weeks in addition to weekly drug and risk reduction counseling for 12 weeks, and then every 4 weeks through Week 52
  Interventions: Drug: Buprenorphine/Naloxone
- Short term medication assisted treatment (ST-MAT) (Experimental): Participants will receive short-term BUP/NX; dosage and length of treatment will be determined by the investigator.Additionally, participants will undergo weekly drug and risk reduction counseling for 12 weeks, and then every 4 weeks through Week 52.
  Interventions: Drug: Buprenorphine/Naloxone

INTERVENTIONS:
Drug: Buprenorphine/Naloxone — Oral tablet
  Other Names: BUP/NX

SUMMARY:
Drug abuse and HIV/AIDS are serious global health problems. Injection drug use is currently the major mode of transmission of HIV in many countries. The purpose of this study is to determine the effectiveness of drug and risk reduction counseling combined with either substitution drug treatment with buprenorphine/naloxone (BUP/NX) or short-term detoxification with BUP/NX in preventing HIV transmission among injection drug users. Participants will be recruited for this study in China and Thailand.

DETAILED DESCRIPTION:
Effective HIV prevention among injection drug users (IDUs) requires educating the at-risk population about HIV transmission and risky behavior, and providing the means for behavior change. Current treatment for opiate dependence focuses on reducing the frequency of drug use. BUP/NX is a combination pill currently used to treat opiate-dependent individuals. This trial will evaluate the effectiveness of two therapies in preventing HIV transmission among IDUs. Drug and risk reduction counseling combined with either long term medication assisted treatment (LT-MAT) with BUP/NX or short term medication assisted treatment (ST-MAT) with BUP/NX will be compared in preventing the transmission of HIV among opiate-dependent individuals.

This study will last 4.5 years. Participants in this study will be randomly assigned to one of two treatment arms. Group 1 will receive LT-MAT with BUP/NX. Group 2 will receive ST-MAT with BUP/NX. An initial 4-week safety and feasibility phase will involve the first 50 participants at each site and will last approximately 30 weeks. Study visits will occur every week and will include a physical exam and blood and urine collection.

The main treatment phase of the study will last 52 weeks. Participants in Group 1 will receive BUP/NX under the tongue, at first daily and then three times a week for 52 weeks. Participants assigned to Group 1 will take part in a BUP/NX reduction phase, which will occur between Weeks 47 and 52. Participants in Group 2 will receive short-term BUP/NX; dosage and length of treatment will be determined by the investigator. Participants assigned to Group 2 will receive BUP/NX for a maximum of 18 days; detoxification may be repeated at Week 26 if the participant is still injecting opiates. After Week 4 of the safety phase and Weeks 26 and 52 of the overall study, participants will complete an intervention acceptability assessment.

In addition, participants in both groups will attend drug and risk reduction counseling weekly. After the first 12 weeks, participants will return every 4 weeks for 10 more counseling sessions. HIV testing, hepatitis C testing, risk assessment, and urine tests for opiates will occur at screening and at Weeks 26, 52, 78, 104, 130 and 156. Plasma from blood samples will be stored at each of these visits. Hepatitis B testing will occur at Week 26. Participants in China will attend study visits through approximately Week 104, and participants in Thailand will attend study visits through approximately Week 156.

Participants in China who have been incarcerated may participate in an optional substudy, which is examining the withdrawal effects from BUP/NX after incarceration. Participants who agree to take part in the substudy will attend one study visit and will complete a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected within 28 days of enrollment
* Meets DSM-IV criteria for opiate dependence
* Positive urine test for opiates
* Injected opiates at least 12 times in the 28 days prior to enrollment, according to self-report
* Willing to use acceptable forms of contraception for the first 12 months of the study
* Able to provide contact information and willing to be contacted by study staff as necessary
* Available for study visits for at least 2 years

Exclusion Criteria:

* Current treatment with methadone, morphine, levo-alpha-acetyl-methadol (LAAM), naltrexone, or nalmefene
* Currently enrolled in another HIV prevention or drug use intervention study
* Known sensitivity to buprenorphine or naloxone
* Requires immediate medical attention for dependence on alcohol, benzodiazepines, or other substances. People who are dependent on tobacco are not excluded.
* Currently injecting drugs of abuse other than opiates, more than twice in the last 28 days, according to self-report
* Psychological disturbance or cognitive impairment that may interfere with the study
* Acute or chronic kidney failure
* Certain abnormal laboratory values
* Any other medical or psychiatric condition that, in the opinion of the investigator, would make participation in this study unsafe
* Pregnant or breastfeeding

Inclusion Criteria for Substudy:

* Current or former participant in HPTN 058 study in Xinjiang who was actively in the long-term treatment arm on stable maintenance dose of Suboxone when detained/arrested (last dose within 2 days of incarceration), resulting in immediate cessation of Suboxone without tapering
* Currently released from detention
* Willing to complete one-time questionnaire
* Willing to sign informed consent

Exclusion Criteria for Substudy:

* Any medical or psychiatric condition that, in the opinion of the investigator, would make participation in the study unsafe, or would otherwise interfere with the study objectives or interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1251 (Actual)
Dates: Start 2008-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Metzger, PhD, Study Chair — Center for Studies of Addiction, University of Pennsylvania
Locations (4):
- China (3):
  - Heng County Ctr. for Disease Control & Prevention CRS, Hengzhou Town, Guangxi
  - Guangxi Ctrs. for Disease Control & Prevention and for HIV/AIDS Prevention & Control CRS, Nanning, Guangxi
  - Xinjiang CRS, Ürümqi, Xinjiang
- CMU HIV Prevention CRS, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aceijas C, Stimson GV, Hickman M, Rhodes T; United Nations Reference Group on HIV/AIDS Prevention and Care among IDU in Developing and Transitional Countries. Global overview of injecting drug use and HIV infection among injecting drug users. AIDS. 2004 Nov 19;18(17):2295-303. doi: 10.1097/00002030-200411190-00010. PMID 15577542
- [Background] Gowing L, Farrell M, Bornemann R, Ali R. Substitution treatment of injecting opioid users for prevention of HIV infection. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD004145. doi: 10.1002/14651858.CD004145.pub2. PMID 15495080
- [Background] Koester S, Glanz J, Baron A. Drug sharing among heroin networks: implications for HIV and hepatitis B and C prevention. AIDS Behav. 2005 Mar;9(1):27-39. doi: 10.1007/s10461-005-1679-y. PMID 15812611
- [Background] Raisch DW, Fye CL, Boardman KD, Sather MR. Opioid dependence treatment, including buprenorphine/naloxone. Ann Pharmacother. 2002 Feb;36(2):312-21. doi: 10.1345/aph.10421. PMID 11847954
- [Background] Ruan Y, Qin G, Liu S, Qian H, Zhang L, Zhou F, He Y, Chen K, Yin L, Chen X, Hao Q, Xing H, Song Y, Wang Y, Hong K, Chen J, Shao Y. HIV incidence and factors contributed to retention in a 12-month follow-up study of injection drug users in Sichuan Province, China. J Acquir Immune Defic Syndr. 2005 Aug 1;39(4):459-63. doi: 10.1097/01.qai.0000152398.47025.0f. PMID 16010170
- [Derived] Lucas GM, Beauchamp G, Aramrattana A, Shao Y, Liu W, Fu L, Jackson JB, Celentano DD, Richardson P, Metzger D; HPTN 058 study group. Short-term safety of buprenorphine/naloxone in HIV-seronegative opioid-dependent Chinese and Thai drug injectors enrolled in HIV Prevention Trials Network 058. Int J Drug Policy. 2012 Mar;23(2):162-5. doi: 10.1016/j.drugpo.2011.06.005. Epub 2011 Aug 17. PMID 21852093
- [Derived] Sugarman J, Corneli A, Donnell D, Liu TY, Rose S, Celentano D, Jackson B, Aramrattana A, Wei L, Shao Y, Liping F, Baoling R, Dye B, Metzger D. Are there adverse consequences of quizzing during informed consent for HIV research? J Med Ethics. 2011 Nov;37(11):693-7. doi: 10.1136/jme.2011.042358. Epub 2011 Jun 8. PMID 21653649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sites were selected based on prior HIV incidence rates among opiate injectors.
  At the first scheduled interim analyses, when 25% of the participants had completed 104 weeks on study, the Data Safety Monitoring Board (DSMB) halted the study due to futility as a result of lower than anticipated HIV incidence rates.
Pre-assignment Details: The study represented the first use of buprenorphine-naloxone as a treatment for opiate dependence in each community, thus implementation of the study and recruitment of participants included a significant effort devoted to community engagement and education. Each site had an active community advisory board (CAB).
Period: Overall Study
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT)
Started | 623 | 628 (1 excluded from analysis (enrollment date exceeded eligibility window by 13 days))
Week 8 | 510 | 443
Week 26 | 460 | 440
Week 52 | 362 | 340
Week 78 | 283 | 285
Visit 104 | 211 | 204
Completed | 211 | 204
Not Completed | 412 | 424
Not completed — Data Safety Monitoring Board (DSMB) halt | 412 | 424

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT) | Total
Number analyzed (Participants) | 623 | 627 | 1250
Age, Customized [Median (Inter-Quartile Range); unit: years] | 33 [27 to 39] | 34 [28 to 39] | 34 [28 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 50 | 99
  Male | 574 | 577 | 1151
Region of Enrollment [Number; unit: participants]
  China | 522 | 527 | 1049
  Thailand | 101 | 100 | 201
Years of Injection [Median (Inter-Quartile Range); unit: Years] | 7 [3 to 12] | 7 [3 to 12] | 7 [3 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Evidence of HIV-1 Infection or Death for Visits up to 104 Weeks
Description: The primary endpoint for the study was cumulative HIV infection or death after a second year of follow-up (i.e. at week 104), one year after completion of the treatment phase, designed to test a durable intervention effect.
Time Frame: For visits up to week 104
Population: Data Safety Monitoring Board (DSMB) halted the study on October 4, 2011 due to futility as a result of lower than anticipated HIV incidence rates. See participant flow section for the number of participants who completed visit up to 104 by July 31, 2012.
Measure: Number; unit: participants
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT)
Number analyzed (Participants) | 477 | 470
participants
  # of HIV infections | 2 | 5
  # of Deaths | 8 | 9
Statistical Analysis 1: Comparison: Long Term Medication Assisted Treatment (LT-MAT); Test type: Superiority or Other; Incident rate per 100 person-years = 1.5, 95% CI 2-sided [0.7 to 2.8]
Statistical Analysis 2: Comparison: Short Term Medication Assisted Treatment (ST-MAT); Test type: Superiority or Other; Incident rate per 100 person-years = 2.2, 95% CI 2-sided [1.2 to 3.7]
Statistical Analysis 3: Comparison: Long Term Medication Assisted Treatment (LT-MAT) vs Short Term Medication Assisted Treatment (ST-MAT); Test type: Superiority or Other; p = 0.3769, Regression, Cox; Cox Proportional Hazard = 0.694, 95% CI 2-sided [0.308 to 1.562]

2. Secondary Outcome: Number of Participants With Urinalysis Results Positive for Opiates
Description: Urine drug screen were assessed monthly and semiannually.
Time Frame: Measured through Week 104
Population: Number of participants presented here applies to visit 104 for whom data available.
Measure: Number; unit: participants
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT)
Number analyzed (Participants) | 208 | 202
participants | 138 | 141
Statistical Analysis 1: Comparison: Long Term Medication Assisted Treatment (LT-MAT) vs Short Term Medication Assisted Treatment (ST-MAT); Test type: Superiority or Other; p = 0.4325, Regression, Logistic — P value applies for the comparison at visit 104; adjusted for site; Odds Ratio (OR) = 0.844, 95% CI 2-sided [0.553 to 1.289]

3. Secondary Outcome: Self-report of Continued Injection Opiate Use in the Last 30 Days
Description: All participants completed interviewer-administered assessments of injection and non-injection drug use at baseline and at semi-annual visits.
Time Frame: Measured through Week 104
Population: Number of participants presented here applies to whom data available at week 104.
Measure: Number; unit: participants
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT)
Number analyzed (Participants) | 208 | 202
participants | 102 | 107
Statistical Analysis 1: Comparison: Long Term Medication Assisted Treatment (LT-MAT) vs Short Term Medication Assisted Treatment (ST-MAT); Test type: Superiority or Other; p = 0.2749, Regression, Logistic — P value applies for the comparison at visit 104 only; Odds Ratio (OR) = 0.800, 95% CI 2-sided [0.536 to 1.194]

4. Secondary Outcome: Number of Participants Reported Using Injection Equipment (Needles, Syringes, Cookers, Cottons, and Rinse Water) in the Prior 6 Months
Time Frame: Measured through Week 104
Population: Number of participants presented here applies to whom data available at week 104.
Measure: Number; unit: participants
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT)
Number analyzed (Participants) | 208 | 202
participants | 23 | 28
Statistical Analysis 1: Comparison: Long Term Medication Assisted Treatment (LT-MAT) vs Short Term Medication Assisted Treatment (ST-MAT); Test type: Superiority or Other; p = 0.3446, Regression, Logistic — Analysis is done for visit 104; Adjusted for site; Odds Ratio (OR) = 0.746, 95% CI 2-sided [0.407 to 1.369]

5. Secondary Outcome: Self-reported Number of Injections in the Last Month
Time Frame: Measured through Week 104
Population: Number of participants presented here applies to whom data available at week 104.
Measure: Median (Inter-Quartile Range); unit: injections
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT)
Number analyzed (Participants) | 623 | 627
injections | 30 [6 to 60] | 30 [7 to 60]
Statistical Analysis 1: Comparison: Long Term Medication Assisted Treatment (LT-MAT) vs Short Term Medication Assisted Treatment (ST-MAT); Test type: Superiority or Other; p = 0.3620, Generalized linear model — P value applies for the comparison at visit 104 only. See the estimation comments for the other visits; adjusted for site; Odds Ratio (OR) = 0.8712, 95% CI 2-sided [0.6477 to 1.1718]

6. Secondary Outcome: Incident Hepatitis C Infections for Thailand and China
Description: HCV antibody using two different HCV EIA assays (Ortho HCV antibody version 3.0 and Wantai HCV antibody assay) at baseline and between 26-156 weeks later.
  If both HCV EIA antibody assays were nonreactive, then the participant was considered not to be HCV infected. If either assay was reactive, then the Ortho HCV assay was repeated in duplicate. If two of 3 Ortho HCV assays were reactive, then the participant was considered to be HCV infected. Samples that were repeatedly reactive for HCV antibody at a follow-up visit were tested for HCV RNA by the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV assay. Not all participants had follow-up testing performed in China due to early closure of the study by the Data Safety Monitoring Board on account of futility due to a low HIV incidence (the primary study endpoint).
  Analysis was done separately for both countries
Time Frame: Measured through week 156 in Thailand and 104 weeks in China
Population: Baseline HCV antibody negative participants.
Measure: Number; unit: participants with HCV antibody
Groups:
- China; Thailand: Long Term and Short arms were compared
Arm/Group | China | Thailand
Number analyzed (Participants) | 132 | 78
participants with HCV antibody | 41 | 8
Statistical Analysis 1: Comparison: China; Test type: Superiority or Other; Incident rate of 100 person-years = 22, 95% CI 2-sided [14.7 to 31.6] — 29 events over 132 person-years
Statistical Analysis 2: Comparison: Thailand; Test type: Superiority or Other; Incident rate of 100 person-years = 4.59, 95% CI 2-sided [2.0 to 9.0] — 8 events over 174 person-years

7. Secondary Outcome: Incident Hepatitis B Infections
Description: Serum samples were tested at baseline and between 26-52 weeks later for Hepatitis B surface antigen (HBsAg) using a commercial enzyme immunoassay (EIA) (Abbott Murex HBsAg version 3.0). If the HBsAg test was initially non-reactive, then the participant was considered to be negative for HBsAg. If the HBsAg test was initially reactive, then it was repeated in duplicate. If at least two of 3 tests were reactive, then the participant was considered to be positive for HBsAg.
Time Frame: Measured through week 52
Measure: Number; unit: participants with HBsAg
Arm/Group | China | Thailand
Number analyzed (Participants) | 607 | 55
participants with HBsAg | 9 | 0
Statistical Analysis 1: Comparison: China; Test type: Superiority or Other; Incident rate of 100 person-years = 2.7, 95% CI 2-sided [1.22 to 5.08] — 9 events over 336 person-years
Statistical Analysis 2: Comparison: Thailand; Test type: Superiority or Other; Incident rate of 100 person-years = 0.0, 95% CI 2-sided [0.00 to 10.1] — 0 events over 37 person-years

ADVERSE EVENTS:
Arm/Group | Long Term Medication Assisted Treatment (LT-MAT) | Short Term Medication Assisted Treatment (ST-MAT)
Serious Adverse Events (participants affected / at risk) | 38/623 | 42/628
Other Adverse Events (participants affected / at risk) | 0/623 | 1/628
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term Medication Assisted Treatment (LT-MAT) (N=623) | Short Term Medication Assisted Treatment (ST-MAT) (N=628)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 1 (1)
Drowning (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bone tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Neurocysticercosis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Penicilliosis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (12) | 14 (14)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vascular rupture (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long Term Medication Assisted Treatment (LT-MAT) (N=623) | Short Term Medication Assisted Treatment (ST-MAT) (N=628)
chest Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study abstracts and publications are subject to HPTN Publication and Public Information Policies and Clinical Trial Agreements between NIAID (DAIDS) and company collaborators. The publication or other disclosure can be delayed for up to thirty additional business days for manuscripts & five business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.